CLINICAL TRIAL: NCT02376829
Title: Class II Correction Study Using the Invisalign System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Align Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRF-002
Record Dates: First submitted 2015-02-11; First posted 2015-03-03 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Malocclusion
Keywords: Orthodontic; Orthodontic Treatment; Clear Aligners; Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- The Invisalign System (Experimental): Class II correction of malocclusions
  Interventions: Device: Invisalign System

INTERVENTIONS:
Device: Invisalign System — The Invisalign® System is indicated for the alignment of teeth during orthodontic treatment of malocclusion

SUMMARY:
To demonstrate that growing teenagers which present up to full cusp Class II malocclusions can be treated using the Invisalign System.

DETAILED DESCRIPTION:
The Invisalign® System consists of a series of clear plastic aligners that are intended to replace conventional wire and bracket technology for many orthodontic cases. Each custom manufactured aligner exerts gentle, continuous forces to move teeth incrementally from their original state to a final, treated state. Each aligner is worn for about two weeks, then replaced by the next in the series until the final position is achieved. For years, orthodontists and dentists have used removable appliances for orthodontic treatment. Today, with the application of computer technology and custom manufacturing, Invisalign treats a broader range of cases with greater precision.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have fully erupted dentition excluding 2nd and 3rd molars
* Age range 11-19 years old
* Subject that requires bilateral Class II correction and must require at least 3mm of correction as measured by first molar relationship

Exclusion Criteria:

* Subject who has unerupted, erupting, partially erupted dentition (except for 2nd and 3rd molars)
* Subject who has spaces between adjacent teeth larger than 3mm
* Subject with active caries
* Subject with periodontal disease
* Subject does not have at least 1st molar fully captured in PVS (polyvinyl siloxane material ) impression or intraoral scan.
* Subject with TMD (Temporomandibular joint dysfunction) symptoms
* Subject has undergone pre-treatment with any orthodontic appliance (any previous treatment prior to study)
* Subject has known allergy to latex and plastic
* Subjects who are pregnant or will become pregnant during treatment

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 164 (Actual)
Dates: Start 2015-03; Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Wilson-Lopes, Study Director — Align Technology, Inc.
Locations (10):
- United States (8):
  - Dr. Gary Brigham, Scottsdale, Arizona
  - Dr. Donna Galante, Rocklin, California
  - Dr. Mark Holt, Roseville, California
  - Dr. Ray Kubisch and Dr. Drew Ferris, Santa Barbara, California
  - Dr. Sandra Selnick, Ellicott City, Maryland
  - Dr. Regina Blevins, Inver Grove Heights, Minnesota
  - Dr. William Kottemann, Maple Grove, Minnesota
  - Dr. Barry Glaser, Cortlandt Manor, New York
- Canada (2):
  - Dr. Sam Daher, Vancouver, British Columbia
  - Dr. Sandra Tai, Vancouver, British Columbia

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinical Study: There were a total of nine (9) Investigators participating in the Clinical Study, seven (7) in the US and two (2) in Canada.
- Continued Access: There were a total of seven (7) Investigators participating in the Continued Access Study, five (5) in the US and two (2) in Canada.
Period: Overall Study
Arm/Group | Clinical Study | Continued Access
Started | 81 | 83
Completed | 54 | 39
Not Completed | 27 | 44
Not completed — Withdrawal by Subject | 27 | 44

BASELINE CHARACTERISTICS:
Population: Race and Ethnicity was not captured as part of this study.
Groups:
- Clinical Study: There were a total of nine (9) Investigators participating in the Clinical Study, seven (7) in the US and two (2) in Canada. All US Investigators have completed their study participation and have been closed out with the Sponsor and the IRB. Both sites in Canada have completed their study participation and have been closed out with the Sponsor and the IRB.
- Continued Access: There were a total of seven (7) Investigators participating in the Continued Access Study, five (5) in the US and two (2) in Canada. As of November 23, 2021, Aall five (5) US Investigators havedve completed their study participation and have been closed with the Sponsor and with the IRB. Both These closed Investigators are: Dr. William Kottemann, Dr. Donna Galante, Dr. Sandra Selnick, Dr. Regina Blevins, and Dr. Raymond Kubisch. As of November 19, 2021, both sites in Canada were closed with the Sponsor and the IRB.
- Total: Total of all reporting groups
Arm/Group | Clinical Study | Continued Access | Total
Number analyzed (Participants) | 81 | 83 | 164
Age, Continuous [Mean (Full Range); unit: Years] | 13.24 [12.59 to 15.28] | 13.17 [12.87 to 16.10] | 13.2 [12.59 to 16.10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 47 | 90
  Male | 38 | 36 | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Rate of Tooth Movement at the End of Class II Correction.
Description: The primary objective will be met through demonstrating that the velocity of Invisalign with MRF overjet correction is non-inferior to the published rates of Dynamax (0.42mm/month).
Time Frame: End of Class II Correction up to 18 months
Population: 1. The Continued Access study was created to be able to offer additional Invisalign with Mandibular Advancement to doctors in the Clinical Study after recruitment had completed. The data has been combined for the primary and secondary objectives for pooling and analysis of the data. The data has been provided to FDA to support the IDE and has been 510K cleared for this device.
Measure: Mean (80% Confidence Interval); unit: mm/month
Groups:
- Primary Objective: The primary objective will be met by demonstrating that the velocity of Invisalign with MRF overjet correction is non-inferior to the published rates of Dynamax (0.42mm/month)3.
Arm/Group | Primary Objective
Number analyzed (Participants) | 42
mm/month | .44 [.37 to .51]

2. Secondary Outcome: Length of Treatment Time
Description: This is the total treatment length of time that subjects took (in days) to complete Invisalign system treatment
Time Frame: End of Treatment approximately 2 years
Measure: Mean (80% Confidence Interval); unit: Days
Groups:
- Secondary Objective: Length of Treatment Time: The secondary endpoints will be measured by evaluating subjects length of treatment time during their Invisalign System treatment.
Arm/Group | Secondary Objective: Length of Treatment Time
Number analyzed (Participants) | 78
Days | 461 [434 to 489]

3. Secondary Outcome: Patient Quality of Life Questionnaire Throughout Treatment
Description: As part of the secondary objective, subject perception was assessed through analysis of case report forms. Case report form analysis of the Quality of Life forms was conducted from the subjects in both the Clinical Study and Continued Access Clinical Study. Subjects were asked to rate their orthodontic experience throughout the course of the study, with options 1(very difficult), 2 (difficult), 3 (average), 4 (easy), and 5 (very easy) as the ratings.
Time Frame: End of Treatment approximately 2 years
Population: The number of participants analyzed in each row is different due to withdrawal and lost to follow up subjects being removed from the study.
Measure: Mean (80% Confidence Interval); unit: score on a table
Groups:
- Average Rating of Orthodontic Experience From Subject Reported Quality of Life Form: Average Rating of Orthodontic Experience from Subject Reported Quality of Life Form. This includes both the Clinical Study (CS) and Continued Access (CAS) portions of the study.
Arm/Group | Average Rating of Orthodontic Experience From Subject Reported Quality of Life Form
Number analyzed (Participants) | 164
score on a table
  Average Rating of Orthodontic Experience From Subject QOL forms-Initial: number analyzed (Participants) | 144
  Average Rating of Orthodontic Experience From Subject QOL forms-Initial | 4.24 [4.15 to 4.33]
  Average Rating of Orthodontic Experience From Subject QOL forms-End of MA: number analyzed (Participants) | 112
  Average Rating of Orthodontic Experience From Subject QOL forms-End of MA | 4.28 [4.18 to 4.38]
  Average Rating of Orthodontic Experience From Subject QOL forms-End of Treatment: number analyzed (Participants) | 84
  Average Rating of Orthodontic Experience From Subject QOL forms-End of Treatment | 4.39 [4.28 to 4.50]

4. Secondary Outcome: Doctor Survey for Satisfaction With Treatment Outcomes
Description: Doctors filled out a Doctor Survey with a scale rating of 1 (very difficult) to 5 (very easy) on how easy the product was to use and their satisfaction with the product. A higher score on the scale meant a better satisfaction experience .
Time Frame: End of Treatment approximately 2 years
Population: The average rating of doctor satisfaction with the subject's treatment outcomes, on a scale of 1 (unsatisfied) to 5 (satisfied).
Measure: Mean (80% Confidence Interval); unit: score on a scale
Groups:
- Doctor Satisfaction With Subject's Treatment Outcome: Rating of Doctor Satisfaction with Subject's Treatment Outcome
Arm/Group | Doctor Satisfaction With Subject's Treatment Outcome
Number analyzed (Participants) | 94
score on a scale | 4.56 [4.45 to 4.67]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of Invisalign System Treatment for each subject for the duration of the study. Adverse Events were monitored through study completion, an average of 2 years.
Description: The definitions for adverse events and serious adverse events for the Invisalign System with Mandibular Advancement Feature are described in the Clinical Study Protocol
Arm/Group | The Invisalign System
All-Cause Mortality (participants affected / at risk) | 0/164
Serious Adverse Events (participants affected / at risk) | 0/164
Other Adverse Events (participants affected / at risk) | 0/164

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT02376829/Prot_SAP_000.pdf